CLINICAL TRIAL: NCT05461391
Title: The Effects of COVID-19 Infection on Respiratory Muscle Strength and Core Stabilization in Healthy Individuals Who Exercise Regularly
Brief Title: The Effects of COVID-19 Infection on Respiratory Muscle Strength and Core Stabilization
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, İldeniz Yalnız, Physiotherapist, Yeditepe University
Other Study IDs: yeditepe123
Record Dates: First submitted 2022-02-12; First posted 2022-07-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Pandemic, COVID-19; Corona Virus Infection
Keywords: covid-19; coronavirus; respiratory physiotherapy; core stabilization
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Participants who got COVID-19.
- Control Group: Healthy participants

SUMMARY:
World Health Organization (WHO) Novel-19 Corrosion Disease (COVID) in 2019 without being used by a pathway caused by the SARS-CoV-2 virus. After the acute period in COVID-19 patients, muscle weakness may continue in breathing, weakness, and training. The effects on core stabilization, pulmonary functions, respiratory muscle strength, physical activity scores and quality of life in healthy adults who do not have COVID-19 who do regular exercise may be higher than in healthy adults who do regular exercise with COVID-19.

DETAILED DESCRIPTION:
The type of our study was planned as Case-Control. 50 exercises will be included in our study. The first COVID-19 (n= 25) is healthy, and the second group will come from the successful group without COVID-19 (n=25). Between February and April, a student will accept participating in the clinic at Bezmialem Foundation University. After being informed about it, the attached form will be signed. In addition, participants will be asked to fill in our attached document, including demographic and clinical studies, in a face-to-face interview. All body exercises, breathing muscle test, six-minute walking test, McGill core endurance test, short-form test, and quality of life test were planned in our two groups. The results of these tests will be evaluated by testing and checking.

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 18-50,
2. Volunteering to participate in the research,
3. Those who have done aerobic exercise at least three days a week in the last three months

Exclusion Criteria:

1. Neurological deficits in the upper or lower extremities,
2. Fractures or orthopedic problems in the upper or lower extremities,
3. Cardiovascular diseases that prevent rehabilitation,
4. Systematic rheumatic disease (rheumatoid arthritis, ankylosing spondylitis),
5. History of surgery in the last three months,
6. Patients with spine problems,
7. Smokers,
8. Patients with chronic respiratory problems.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Data will be evaluated in healthy adult volunteers who agreed to participate in the clinical study at Bezmialem Vakıf University Dragos Hospital between February and April.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test | 8 weeks
  Medical International Research Spirodoc® Spiro spirometry will evaluate the respiratory functions of Italian brand volunteers. Lung function tests can determine both expected values and deviations of lung volumes. Spirometry has been used for over 150 years. Spirometry tests objectively evaluate both inspiratory and expiratory patients. The test will be repeated three times, and the best values will be recorded before and after the interventions.
Respiratory Muscle Strength | 8 weeks
  Mikro Medical Micro RPM is aimed to measure Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) values. During the application, maximum effort is requested, and the patient will be shown the test beforehand. During the measurement of MIP and MEP, it is closed with a nose clip, and after a deep breath, volunteers will be asked to give a maximum exhale for 1 to 3 seconds.
Six Minute Walk Test (6MWT) | 8 weeks
  The 6MWT is a test that patients most commonly use, is valid, inexpensive, popular, easy to tolerate, easy to use, has minimal technological resources, and shows daily activity compared to other walking tests. They will be asked to walk at the same speed for 6 minutes, but not to run, on a 30-meter straight corridor. The volunteers' distance walked in 6 minutes will be calculated and evaluated.
McGill Core Endurance Test | 8 weeks
  McGill Core Endurance Test consists of 4 different test positions. It assesses the core endurance of volunteers.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | 8 weeks
  The IPAQ is the most widely used physical activity questionnaire to describe young and middle-aged adults (15-69 years) participation in physical activity. IPAQ-SF (short form) provides individual results for walking, moderate-intensity, and vigorous-intensity activity scores. The three physical activities' duration (in minutes) and frequency (in days) give the total score. Scores used for Mean Metabolic Task Equivalent (MET) values, total physical activity MET-minutes/week = Total walking + Moderate + Vigorous MET minutes/week scores. Survey questions will be asked to the participants face to face by the researcher, and the answers will be recorded.
Quality of Life Scale (SF36) | 8 weeks
  It was planned to evaluate the quality of life of the volunteers with SF36.
Dyspnea Scale | 8 weeks
  The Modified Medical Research Council Scale (MMRC) is used to investigate the severity of dyspnea during activity in people with and without the disease. The MMRC is a five-item scale based on various activities that cause shortness of breath. Volunteers easily mark the activity level that causes dyspnea on the scale. The story of dyspnea in patients is graded from the "0" point, and the "0" point indicates the absence of dyspnea. The survey questions will be asked to the participants face to face by the researcher, and the answers will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ildeniz yalnız, Study Director — Bezmialem Vakif University Dragos Hospital; elif develi, Principal Investigator — Yeditepe University
Locations (1):
- Bezmialem Vakif University Dragos Hospital, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiumello D, Coppola S, Froio S, Gotti M. What's Next After ARDS: Long-Term Outcomes. Respir Care. 2016 May;61(5):689-99. doi: 10.4187/respcare.04644. PMID 27121623
- [Background] Cavaggioni L, Ongaro L, Zannin E, Iaia FM, Alberti G. Effects of different core exercises on respiratory parameters and abdominal strength. J Phys Ther Sci. 2015 Oct;27(10):3249-53. doi: 10.1589/jpts.27.3249. Epub 2015 Oct 30. PMID 26644685
- [Background] The Novel Coronavirus Pneumonia Emergency Response Epidemiology Team. The Epidemiological Characteristics of an Outbreak of 2019 Novel Coronavirus Diseases (COVID-19) - China, 2020. China CDC Wkly. 2020 Feb 21;2(8):113-122. No abstract available. PMID 34594836
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Chhabra SK. Clinical application of spirometry in asthma: Why, when and how often? Lung India. 2015 Nov-Dec;32(6):635-7. doi: 10.4103/0970-2113.168139. No abstract available. PMID 26664177
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] FLETCHER CM. The clinical diagnosis of pulmonary emphysema; an experimental study. Proc R Soc Med. 1952 Sep;45(9):577-84. No abstract available. PMID 13003946
- [Result] Develi E, Subasi F, Aslan GK, Bingol Z. The effects of core stabilization training on dynamic balance and pulmonary parameters in patients with asthma. J Back Musculoskelet Rehabil. 2021;34(4):639-648. doi: 10.3233/BMR-191803. PMID 33720873

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT05461391/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT05461391/SAP_001.pdf